CLINICAL TRIAL: NCT01180010
Title: Low-Dose Chest CT for Lung Cancer Screening in Survivors of Hodgkin's Disease
Brief Title: Low Dose Chest Computed Tomography (CT) Screening
Status: Completed | Type: Observational
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Other Study IDs: UHN REB 08-0294-CE
Record Dates: First submitted 2010-08-10; First posted 2010-08-11 (Estimated); Last update posted 2016-12-29 (Estimated); Status verified 2016-12

CONDITIONS: Hodgkin's Lymphoma
Keywords: Hodgkin's Lymphoma; Lung Cancer; Lung Nodule; CT scan
MeSH Terms: conditions — Hodgkin Disease; Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Procedure: Low Dose CT — A chest CT uses special radiographic equipment using x-rays to capture images of the chest, and with the aid of a computer, processes the images to create cross-sectional pictures or "slices" of the areas of interest. The images can then be printed out or examined on a monitor. The CT scanner is a large unit with a hole running directly through its center, giving the appearance of a doughnut. During the scanning, patients will lie flat on their back on a table, and they are periodically asked to hold their breath. The table will first move through the scanner to determine the correct starting position. The rest of the scans are made as the table moves more slowly through the cavity in the scanner.

SUMMARY:
This research study is being done because patients with a history of chest radiation treatment for Hodgkin's disease have been shown to be at increased risk for developing lung cancer a number of years out from treatment. The risk appears to be further increased among patients with a smoking history. In this study, the CT scans will be read and interpreted by the study radiologist, and the results recorded in a consistent manner. Depending on the findings of the initial CT scan, we will then either repeat the scan in 1 year, or if indicated, send you for further scans or a biopsy. The information collected in this study will help researchers and clinicians in providing more concrete recommendations and screening guidelines for future survivors of Hodgkin's disease who have had similar exposures to radiation and/or chemotherapy and smoking.

ELIGIBILITY:
Inclusion Criteria:

1. 5 years or longer from initial Hodgkin's disease diagnosis
2. Current age 18 or older
3. Received mediastinal irradiation and/or alkylating-agent based chemotherapy
4. Smoking history of 10-pack years or more, or current smoker

Exclusion Criteria:

1. Patients with a history of lung cancer
2. Patients currently receiving treatment for another cancer diagnosis (patients with another cancer, but currently disease-free and not receiving treatment are eligible)
3. Patients with known diagnosis of any metastatic cancer
4. Pregnant women. Female patients must: be at least one year post-menopausal, have had a hysterectomy, or have a serum pregnancy test to confirm that they are not pregnant. These measures must be taken in order to avoid doing a CT scan of a pregnant woman.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for Hodgkin's Lymphoma
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2010-08; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Lung cancer detection rate using chest CT screening in patients at increased risk of lung cancer after Hodgkin's disease therapy. | 5 years
False-positive rates of using chest CT for lung cancer screening in this population. | 5 years

SECONDARY OUTCOMES:
The stage distribution, clinical characteristics and pathologic features of the detected lung cancer | 5 years
The treatment and treatment outcome of lung cancer after Hodgkin's disease in a cohort of patients undergoing routine chest CT screening | 5 years

CONTACTS AND LOCATIONS:
Overall Officials: David Hodgson, MD, Principal Investigator — University Health Network, Princess Margaret Hospital
Locations (1):
- University Health Network, Princess Margaret Hospital, Toronto, Ontario, Canada